CLINICAL TRIAL: NCT03216785
Title: Cohort Study of Patients Patients in the Medical Intensive Care Unit to Evaluate Postintensive Care Sydnrome
Brief Title: SNUH MICU Cohort Study of PICS
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Assistant Professor, Seoul National University Hospital
Other Study IDs: 1704140848
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Critical Care; Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective registry of patients admitted to the medical intensive care unit Patients discharged are followed up to 5 years after discharge

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical intensive care unit

Exclusion Criteria:

* Patients admitted to the intensive care unit for simple procedures
* Patients admitted for postoperative care observation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the medical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Functional status | 3 month
  Clinical frailty scale, The de Morton Mobility Index

SECONDARY OUTCOMES:
Survival | 1 year
  Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No